### INFORMATION FOR PATIENTS

TITLE OF STUDY: MDMA-ASSISTED PSYCHOTHERAPY WITH 12 PATIENTS WITH THERAPY-RESISTANT POSTTRAUMATIC STRESS DISORDER (PTSD).

Dear Patient,

#### **OBJECTIVE AND BACKGROUND OF THE STUDY**

This study examines the safety and effectiveness of MDMA-assisted psychotherapy with 12 patients with Posttraumatic Stress Disorder (PTSD).

PTSD is a mental illness, which can develop as a consequence of traumatic, life-threatening events such as sexual violence, accidents, natural disasters, war, torture, etc. Those afflicted suffer from repeated and undesired, acute memories, mental images and feelings from the trauma and try to master these by avoiding 'triggers' and through avoidance behaviour. They also suffer from hyperarousal, which leads to nervousness, concentration and sleep problems. The private and working life of those afflicted by PTSD is often substantially restricted by these symptoms.

MDMA is classified as a narcotic and may be used only within the context of scientific research. MDMA is also known as "Ecstasy" and is illegally misused as a party drug. MDMA has already been examined legally in many scientific studies.

You have been asked whether you would be willing to participate in this study, because you suffer from PTSD, and because your symptoms did not abate after at least one previous treatment.

### **MDMA-ASSISTED PSYCHOTHERAPY**

Earlier investigations and experiences with the use of MDMA in psychotherapy showed that MDMA-assisted psychotherapy can be effective in the processing of the psychological consequences of traumatic experiences. The psychological effect of MDMA manifests as a enhanced mood; easier access to traumatic and painful memories; lessening of fear, of feelings of guilt and of negative self-evaluation; a feeling of closeness and trust to other people; development of new life perspectives and more positive evaluation of past and present life circumstances.

### **DURATION AND PROCEDURES**

Participation in this study will last approximately 4½ months (duration of treatment) and will include at least 17 consultations.

Screening procedure: This takes place 2-3 weeks before the beginning of the study and comprises a physical and psychiatric investigation, urine tests for drugs and (for women of childbearing age) pregnancy test, blood tests, including HIV test (AIDS test) and electrocardiograph. You are also asked about the symptoms of your PTSD and the triggering traumatic experience. Following enrolement to the study, approx. two weeks later an examination takes place, during which the symptoms of your PTSD are assessed, and an electro encephalograph (EEG) recording is made, combined with psychological questionnaires. Further assessments of your PTSD symptoms are made during and after the conclusion of the treatment (3 weeks, 2, 6 and 12 months after the last MDMA session), and another EEG recording is made after the treatment, 3 weeks after the last MDMA session.

During the entire duration of the study (phases 1 and 2, see below) and until 2 months after the last MDMA session, you are not allowed to take any psychopharmacological drugs. The prior taking of psychopharmacological drugs is stopped in good time. You may continue inprogress psychotherapy during the study; however, you must not increase the frequency of

Version 17.12.07

MDMA-ASSISTED Treatment, Phase 1: After 2 preparatory meetings with the therapists, at which you are given exact instructions concerning the course of the study and the rules of conduct, the first MDMA session takes place. You receive either a full dose of MDMA (125 mg followed by 62.5 mg after 2.5 hours) or a low dose (placebo) of MDMA (25 mg followed by 12.5 mg after 2.5 hours). In phase 1 of the study, 8 of the 12 patients receive the full dose and 4 of the 12 patients the low dose of MDMA. The dose remains the same during all 3 MDMA sessions. The allocation is determined in advance and effected according to the random principle. Thus, neither you nor the researchers know whether you receive a low dose or a full dose. The session lasts 6-8 hours, during which time you mostly lie down, follow the MDMA-triggered internal mental process, listen to music, or talk with the therapists. During the treatment process, you are given support by the therapists. You remain overnight at You can have one previously designated person with you to give you support during the evening and night. On the following day, a first discussion of your experiences of the previous day takes place. Over the following 2-4 weeks, 2-4 integrating psychotherapy sessions take place. The two further MDMA sessions take place each after an interval of 3-5 weeks, respectively, with the same number of followup psychotherapy sessions and following the same procedure. A termination session takes place 3 weeks after the third MDMA session. During phase 1, altogether 2 scientific evalutation sessions take place, at which your PTSD symptoms are assessed.

MDMA-ASSISTED Treatment, Phase 2: Test participants, who in phase 1 of the study received a placebo (a low dose of MDMA) and are dissatisfied with the result of the treatment, have the possibility to participate in phase 2. Participation in phase 2 is voluntary. In phase 2 you will undergo once again the same treatment as in phase 1. At the 3 MDMA sessions, however, you will receive the full dose (125 mg followed by 62.5 mg after 2.5 hours). Phase 2 lasts another 3½ months and will include at least 14 consultations. During phase 2, altogether 2 scientific analysis sessions take place.

Additional scientific evaluation sessions: Both, the participants who received the full dose of MDMA, and those who received the placebo, respectively, in phase 1, but do not wish to participate in phase 2, will be asked again concerning their PTSD symptoms 2, 6 and 12 months, respectively, after the end of the last MDMA session of phase 1.

Participants who also go through phase 2, are asked again concerning their PTSD symptoms 2, 6 and 12 months, respectively, after the end of the last MDMA session of phase 2. For exact time schedule please see supplement.

# **MDMA: SIDE EFFECTS**

<u>Frequent:</u> Lack of appetite, muscle tension in the jaw region, dry mouth, disturbance of equilibrium and decrease in concentration.

<u>Less frequent</u>: Feelings of warmth and/or cold, accelerated heart beat, perspiration, feeling of dizziness, tiredness, stomach upset, states of tension, trembling, headaches or a feeling of weakness, slight changes in your seeing or hearing. All these side effects are slight and usually from 2-3 hours up to a maximum of 24 hours. Exceptionally, conditions of tiredness, irritability or exhaustion can occur, which may continue for more than 3 days.

### **MDMA: RISKS**

# Blood pressure and pulse:

MDMA increases the blood pressure and the pulse. The effects on the blood circulation last approx. 4 to 6 hours. With the dosage used in this study, only a moderate increase of blood pressure and pulse frequency is anticipated. For safety's sake, your blood pressure, pulse and temperature are supervised during the MDMA experience.

Anxiety:

States of nervousness or fearfulness can sometimes occur, but normally these last less than 30 minutes. Due to your PTSD, you could also experience more severe states of fear or other unpleasant feelings. If you learn to permit these to occur and accept them, this can have a positive therapeutic effect. If you cannot deal with these experiences, the test manager will help you when you are in that state and, should you still be excited or very afraid after the end of the experimental session, he/she will remain with you and/or give you medicaments.

<u>Serious problems</u>: Serious problems such as high fever, states of confusion caused by excessive intake of fluids, cramps, liver damage or even cases of death, such as have sometimes been observed with illegal and excessive use of MDMA at parties, have not arisen so far in the context of scientific investigations.

<u>Immune reaction</u>: MDMA can cause a discreetly limited immune reaction during 2 or 3 days after ingestion, comparable with the effect of 4 to 5 alcoholic beverages. This means that during this time you have a somewhat increased risk of catching a cold or some other minor infection.

<u>Addiction</u>: The risk of becoming addicted to MDMA is small. A study of persons who received MDMA for the first time during a scientific investigation, showed that later, outside of this investigation, these test subjects did not have a craving for MDMA.

<u>Long term damage</u>: Based on present scientific data, the researchers assume that you will suffer no permanent changes in the brain, no lasting changes in memory performance and no lasting increase of depressive symptoms or states of fear.

<u>Driving:</u> Up to 24 hours after being ingested, MDMA can impair your ability to drive a vehicle. If, within three days, you are tested for MDMA in the context of a traffic check, this test can be positive. You receive a card from the test manager with his telephone numbers and a note stating that you can test positively due to participation in a clinical trial using MDMA.

<u>Women of childbearing age</u>: The effects of MDMA on the unborn child are not known. Therefore, during the entire study and for at least one month after conclusion of the study, women of childbearing age must practice a safe birth control method. They are tested for pregnancy at the beginning of the study and again before each MDMA or placebo session.

#### **POSSIBLE USEFULNESS**

There is no guarantee that your participating in the study will be of use to you. It is anticipated that the treatment with the full dose of MDMA will improve your PTSD symptoms. The knowledge gained through your participation in this study can help to develop a new method of treatment in the future for patients with PTSD.

### **NEW FINDINGS**

If, during your participation in this study, substantially new findings become known into the treatment of PTSD or about the effects of MDMA that are of significance for you and which clearly deviate from the information in this patient information brochure, then the test managers will communicate this knowledge to you.

# OTHER TREATMENT POSSIBILITIES

It is possible that the treatment that you receive during this study cannot improve your PTSD. There is the alternative of rejecting participation in this study and deciding in favour of another method of treatment, such as, for example, CBT (Cognitive Behaviour Therapy), EMDR (Eye Movement Desensitization and Reprocessing), psychodynamic therapy or treatment with medicaments. The test managers can give you more information in this.

### **DATA SECURITY**

In this study, some of your personal data are recorded. These data are subject to the same confidentiality as other medical documents. They are accessible only to specialists for scientific evaluation. Your identity is not thereby revealed. The specialists in charge, the ethics commission, as well as the members of the authorities responsible can view the data within the context of inspections. At all times - during, before and after the study - the strict confidentiality of your data is guaranteed.

Version 17.12.07

### COSTS, PAYMENT FOR PARTICIPATION AND INSURANCE COVER

No costs accrue for you as a result of your participation in this study. The costs of all examinations and treatments during the study are covered by the sponsors. You will not be paid for your participation in this study. Travel expenses are reimbursed as follows: Travel expenses by public transport or the equivalent amount, if you come by car. If the return journey be not possible within the same day, up to per night to cover all hotel bills will be recompensed to you. The sum total shall not amount to more than per study phase (phase 1 and 2).

| MAP | (Multidisciplinary Association for Psychedelic Studies, USA), their representative ii |
|---|---|
| | and the principle investigator, |
| | , will make good any damages that you may suffer in the context of the clinical |
| trial. | |
| То со | ver their own third-party liabilities and those of the principle investigator, |
| | , MAPS has taken out relevant third-party liability insurance cover with |
| insura | ance Company. If you experience health problems or other damage during or after the |
| clinica | al trial, then please contact the physician in charge, least the physician in charge, least the physician in charge, |
| ensur | e that you receive the necessary medical care and that the information will be provide |
| (notifi | ed) to the insurance company. He knows the current legislation and has the relevar |
| writte | n documents. In the case of damage in the context of the trial, he can give you fire |
| inform | nation on how you can assert a valid claim for damages. In case of dispute, jurisdiction |
| shall l | be at the place of your Swiss domicile. |

#### **VOLUNTARY PARTICIPATION**

Your participation in this study is voluntary. If you wish to forgo participation in this study, you need fear no disadvantages - e.g. for some sort of study-independent treatment. The same applies, if you later withdraw your already-given consent. You have this possibility at any time. You do not have to justify a revocation of your consent and/or your withdrawal from the study. In this case, for your security you undergo a final medical examination.

# **EXCLUSION FROM THE STUDY**

The principle investigator, the sponsors, the responsible authorities or the ethics commission, can, at any time, with or without your consent, interrupt the study or exclude you personally from it, for the following reasons: if you show side effects from the MDMA; if you do not keep the appointments; if you do not take the substance as agreed; if you become pregnant; if you test positively for drugs; or if the study is stopped by the authorities or the sponsors.



# Written Declaration of Consent by Participants of a Clinical Trial

- Please read this form carefully.
- Please ask, if there is something you did not understand or would like to know.

# Information regarding the Clinical Trial

Title of Clinical Trial: MDMA-ASSISTED PSYCHOTHERAPY WITH 12 PATIENTS WITH

THERAPY-RESISTANT POSTTRAUMATIC STRESS DISORDER

(PTSD).

Number of Clinical Trial: 2006/026 (EKO-0511)/2006 DR 2157

**Location of Clinical Trial** 

Principle Investigator, surname and first name:

Participant, surname and first name:

Date of Birth:

Sex:

### Declaration

- I have been informed orally and in writing by the undersigned investigator about the goals and the procedure of the clinical trial, the effects that can be expected, the possible advantages and disadvantages, and possible risks.
- Other possible treatments and treatment procedures have been explained to me.
- I have read and understood the written information from 17.12.07 for participants concerning the trial referred to above. My questions in connection with the participation in this clinical trial have been answered to my satisfaction. I shall receive a copy of my written declaration of consent as well as the information for participants.
- I had sufficient time to make my decision.
- I have been informed about the fact that I shall be compensated by the Multidisciplinary Association for Psychedelic Studies (MAPS) for possible injuries that I may suffer in connection with the clinical trial. It was explained to me that for this purpose, Dr.med. Peter Oehen has taken out an insurance cover with Insurance Company.
- I agree that the responsible specialists of MAPS as well as representatives of the health authorities and the ethics commissions may view my medical data for test and control purposes. The confidentiality of these data is strictly guaranteed.
- I am participating voluntarily in this clinical trial. At any time and without giving any reasons I can revoke my agreement to participation in the same, without thereby incurring any disadvantages for myself with regard to further medical care. In this case, I shall undergo a final medical examination for my own safety.
- I am aware of the fact that during the clinical trial the requirements and restrictions specified in the information for participants must be adhered to. In the interest of my health, the principle investigator can exclude me at any time from the clinical trial. In addition, I shall inform the examiner about any simultaneous treatment by another physician and the taking of medicines (whether prescribed by the physician or obtained independently).

Place, date:

Signature of test person

Place, date:

Name of PI in capital letters Signature of PI

Version 17.12.07